CLINICAL TRIAL: NCT05247476
Title: Type 2 Deiodinase Gene Polymorphism and the Treatment of Hypothyroidism Caused
Brief Title: Type 2 Deiodinase Gene Polymorphism and the Treatment of Hypothyroidism Caused by Thyroidectomy in Thyroid Cancer Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-123
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Cancer, Papillary; Hypothyroidism
Keywords: type 2 deiodinase, TSH suppression
MeSH Terms: conditions — Thyroid Cancer, Papillary; Hypothyroidism | interventions — Thyroid (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-T4 therapy group (Active Comparator): Patients with refractory hypothyroidism still receive L-T4 therapy as usual.
  Interventions: Drug: L-T4
- L-T4+T3 therapy group (Experimental): Patients with refractory hypothyroidism receive L-T4+T3 therapy
  Interventions: Drug: L-T4+T3 (thyroid tablet)

INTERVENTIONS:
Drug: L-T4 — Patients with refractory hypothyroidism continued to receive L-T4 therapy. The drug dose was adjusted so that FT4 did not exceed the normal range, and the TSH suppression target was achieved as far as possible.
  Arms: L-T4 therapy group
Drug: L-T4+T3 (thyroid tablet) — Patients with refractory hypothyroidism changed to receive L-T4 +T3 therapy. The drug dose was adjusted so that FT4 did not exceed the normal range, and the TSH suppression target was achieved as far as possible.
  Arms: L-T4+T3 therapy group

SUMMARY:
This project analyzes the relationship between type 2 deiodinase gene polymorphism and the TSH inhibitory treatment efficacy in thyroid cancer patients with thyroidectomy, and explored the factors influencing TSH inhibitory treatment efficacy. It further explores whether patients with diO2-Thr92ALA genotype or DIO2 Orfa-Gly3ASP genotype should choose T4+T3 treatment, and the effect of different treatment options on the quality life of patients.

DETAILED DESCRIPTION:
Object: To explore the relationship between type 2 deiodinase gene polymorphism and the TSH inhibitory treatment efficacy in thyroid cancer patients with thyroidectomy, And figure out if it is better for patients with diO2-Thr92ALA genotype or DIO2 Orfa-Gly3ASP genotype to choose T4+T3 treatment,

Design:

Part I: Analysis of the correlation between DIO2 genotype and TSH inhibitory treatment effect:

1. In accordance with inclusion and exclusion criteria; A total of 100 patients undergoing total thyroidectomy for thyroid cancer and 100 patients receiving 131 iodine treatment after total thyroidectomy will be included in our hospital from October 2021 to October 2022. All the patients signed informed consent
2. Detection of basic condition:

   The included patients were recorded with height, weight, BMI, routine biochemistry, homocysteine, thyroid function, thyroid peroxidase antibodies, thyroglobulin, thyroid globulin,
3. Genotype detection of DIO2 gene RS225014 and RS12885300 loci were tested for all the patients.
4. Regular L-T4 treatment and drug dose adjustment:

   Patients included in the study were treated with L-T4 daily and the drug dose was adjusted so that FT4 did not exceed the normal range, and the TSH inhibition target was achieved as far as possible. After 3 months' treatment. The data of height, weight, BMI, routine biochemistry, thyroid function, thyroid peroxidase antibodies, thyroglobulin, thyroid globulin were tested again. SF-36 health survey were tested to evaluated the living quality.
5. The effect of genotype and allele frequency on TSH inhibitory treatment was analyzed.

Part II: Compare the effects of single L-T4 treatment and L-T4+T3 on TSH inhibitory treatment and side effects

1. L-t4 treatment vs T4+T3 treatment:

   Through the analysis of the first step, patients with refractory hypothyroidism whose FT4 dose reached 1.9ug/kg/d and TSH inhibition treatment failed to reach the standard were screened out, and these patients were randomly divided into L-T4 treatment group and L-T4+T3 treatment group. The patients were followed up for half a year, and the drug dose was adjusted every month to make TSH inhibition treatment target as far as possible.
2. After half a year of treatment, the height, weight, BMI, routine biochemistry, thyroid function, thyroid peroxidase antibody, thyroglobulin, thyroglobulin antibody, were examined again. All patients were reevaluated SF-36 health survey.
3. Statistical analysis was made of the effects of different treatment methods on TSH inhibition therapy and the effects on patients' quality of life,

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Patients with Hypothyroidism after total thyroidectomy for papillary thyroid carcinoma
3. Patients were informed of the study and voluntarily willing to participate.

Exclusion Criteria:

1. Having depression or other mental illness
2. Taking drugs that interfere with thyroid hormone absorption for other chronic diseases
3. impaired liver function, defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
4. impaired renal function ,eGFR: <45 mL/min (calculated by MDRD formula)
5. Recent Cardiovascular Events in a patient:

(1)Acute Coronary Syndrome (ACS) within 2 months prior to enrolment (2).Hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment (3)Acute Stroke or TIA within two months prior to enrolment (4)Less than two months post coronary artery revascularization 6. Congestive heart failure defined as New York Heart Association (NYHA) class IV, unstable or acute congestive heart failure.

7. Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
TSH suppression | Up to 6 months
  The TSH level can reach the aim of the TSH suppresion therapy

SECONDARY OUTCOMES:
quality life evalutaion | Up to 6 months
  evaluate the quality life of the patients with SF-36 survey.

CONTACTS AND LOCATIONS:
Overall Officials: Yilin Zhao, Study Director — Zhongshan Hospital Xiamen University
Locations (1):
- Yan Ling, Xiamen, Fujian, China